CLINICAL TRIAL: NCT02107911
Title: Factors Affecting the Intention to Take Non-occupational HIV Post-exposure Prophylaxis Among Thai Men Who Have Sex With Men
Brief Title: Factors Affecting the Intention to Take nPEP Among Thai MSM
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Responsible Party: Principal Investigator, Nitiya Chomchey, Ms.Nitiya Chomchey, RN, MSc, SEARCH Research Foundation
Other Study IDs: SEARCH 020
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: HIV; Homosexuality
Keywords: men who have sex with men; non-occupational post exposure prophylaxis; HIV infection
MeSH Terms: conditions — Homosexuality; HIV Infections

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- men who have sex with men: MSM who seek voluntary HIV counseling and testing service at the Anonymous Clinic, TRC-ARC, including those who describe risky sexual exposure to HIV within the preceding 72 hours and meet nPEP criteria.

SUMMARY:
The potential participants will be informed of the study details, including the study objectives. Once they have read the study information sheet and have a good understanding of the study, those who intend to participate in the study will be asked to sign the consent form for this study. There are 2 groups of participants: MSM who seek HIV voluntary counseling and testing service (phase I) and MSM who meet nPEP criteria (phase II).

DETAILED DESCRIPTION:
This study design is mixed-method, starting with quantitative research and followed by qualitative research. The study will be conducted in 2 phases: a cross-sectional study during phase I and a prospective descriptive study during phase II, which will use qualitative research techniques to help understand and define obstacles and uncover opportunities to improve adherence to post-exposure prophylaxis.

During phase I, this study is a quantitative research study using a cross-sectional study design which aims to enroll 450 men who have sex with men (MSM) within 6 months and to collect data by administration of questionnaire amongst all MSM via face-to-face interview. During phase II, we will use a quantitative research design and perform in-depth interviews with those MSM who choose to receive and choose not to receive nPEP despite the fact that they meet nPEP criteria. We expect to identify approximately 50 MSM who meet nPEP criteria during the enrollment period. The number of volunteers will be determined based on saturation theory in which the data collection will be considered complete after analysis of the data shows that additional entries provide no further information (64). The number of volunteers in phase II may not be able to be specified with certainty in advance. Enrollment of subjects will stop once data acquisition is saturated.

An initial review of demographic data and sexual behavior amongst MSM seen at the TRC-ARC will be undertaken by interviewing the TRC-ARC staff who are responsible for looking after this population. This process will aid understanding of clinic logistics and help identify opportunities to meet with MSM individuals. The potential participants will be informed of the study details, including the study objectives. Once they have read the study information sheet and have a good understanding of the study, those who intend to participate in the study will be asked to sign the consent form for this study. There are 2 groups of participants: MSM who seek HIV voluntary counseling and testing service (phase I) and MSM who meet nPEP criteria (phase II).

Phase I. MSM who seek HIV voluntary counseling and testing

1. All MSM clients will be interviewed to complete the questionnaires designed to collect information for this study before the pre-test counseling. The questions will collect demographic data and data regarding HIV risk behaviors, HIV knowledge, intention to take nPEP, factors affecting the intention to take nPEP, experience on nPEP use, and awareness of nPEP.
2. After MSM clients receive the counseling. They will be interviewed to answer the questionnaires about HIV knowledge, intention to take nPEP, factor affecting to intention to take nPEP, nPEP knowledge.
3. All MSM clients will receive pre-test counseling, HIV testing, and post-test counseling according to the standard of care at the Anonymous Clinic, TRC-ARC. Counselors will also assess clients for nPEP eligibility criteria according to the standard clinic guidelines.

Phase II. MSM who receive nPEP

1. Participant who describes a history of an HIV risk exposure within the preceding 72 hours and meets nPEP eligibility criteria as assessed by the clinic counselor. After participants receive all information to know whether they receive antiretroviral medication, they can decide by themselves about taking medication. The participant who select to take nPEP will receive a 14-day supply of nPEP medication and will be scheduled back to receive the rest of their medication.
2. Both participant who decide to take and not take nPEP will be asked to take part in the in-depth interviews to examine factors affecting the decision to use nPEP.
3. At week 6, the participants who take nPEP will be evaluated for HIV infection, adherence to medication during the 28-day course of nPEP, side effects from nPEP and asked to be interviewed about risk behaviors and other HIV prevention methods since the start of nPEP.

At each of these study visits, the participant will receive risk reduction counseling along with the provision of condoms and lubricant

In accordance to the standard of care at the Anonymous Clinic, TRC-ARC, participants who decide to take nPEP (whose risk of HIV exposure must be within the preceding 72 hours) will receive 3 antiretroviral medications; 2 nucleoside reverse transcriptase inhibitors plus 1 protease inhibitor or non-nucleoside reverse transcriptase inhibitor. The clients will receive HIV antibody testing prior to taking nPEP and at week 6 after starting nPEP.

ELIGIBILITY:
Phase I

Inclusion criteria:

* Thai MSM seeking HIV voluntary counseling and testing at the Anonymous Clinic, TRC-ARC.
* Age >18 years old.
* Read and understand the study and document their consent on the informed consent form.

Exclusion criteria:

* Any individual who has any medical or psychological conditions, including drug or alcohol addiction that the physician or counselor feels may interfere with his ability to participate in the study or cannot provide adequate information.
* Any MSM who is already receiving antiretroviral therapy for the prevention of HIV infection after exposure to HIV.

Phase II

Inclusion criteria:

* Thai MSM who meet nPEP criteria
* Document their consent on the informed consent form of in-depth interview

Exclusion criteria:

* Cannot come to the clinic according to the schedule visit
* Individual who has any medical or psychological conditions, including drug or alcohol addiction that the investigator feels may interfere with his ability to attend study visits or cannot provide the information

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSM who seek voluntary HIV counseling and testing service at the Thai Red Cross AIDS Research Centre, including those who describe risky sexual exposure to HIV within the preceding 72 hours and meet nPEP criteria.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Intention to take nPEP | 1 day

SECONDARY OUTCOMES:
Knowledge and awareness regarding nPEP | 1 day
Knowledge and awareness about HIV risk behaviors | 1 day
Stigma and discrimination towards HIV | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Nitiya - Chomchey, MSc, Principal Investigator — SEARCH, the Thai Red Cross AIDS Research Centre
Locations (1):
- SEARCH, the Thai Red Cross AIDS Research Centre, Bangkok, Bangkok, Thailand